CLINICAL TRIAL: NCT01679483
Title: THE ROLE OF FLOSEAL IN THE PREVENTION OF LYMPHOCELE AND LYMPHATIC ASCITES AFTER LYMPH NODE DISSECTION FOR GYNECOLOGIC CANCER: A RANDOMIZED CONTROLLED TRIAL
Brief Title: Efficacy Study of FloSeal for Prevention of Lymphocele After Lymphadenectomy for Gynecologic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FloSeal-LND
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Gynecologic Cancer; Cervical Cancer; Endometrial Cancer; Ovarian Cancer; Fallopian Tubal Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FloSeal group (Experimental): This group will undergo appropriate cancer surgery for each patient with pelvic lymph node dissection +/- para-aortic lymph node dissection. At the completion of lymph node dissection, 2 vials of Floseal will be applied to each lymph node area.
  Interventions: Drug: FloSeal application
- No FloSeal group (No Intervention): All surgical procedures of control group is the same with study group except that Floseal is not applicated in control group.

INTERVENTIONS:
Drug: FloSeal application — At the completion of lymph node dissection, 2 vials of Floseal will be applied to each lymph node area.
  Arms: FloSeal group

SUMMARY:
To compare the incidence of lymphocele and lymphatic ascites between patient who use versus who do not use FloSeal during lymph node dissection

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary cancer of the uterine cervix, uterine corpus, ovary, and fallopian tube
* FIGO stage Cervical cancer: FIOG stage IA2-IIA2 Uterine cancer: FIGO stage I-III Ovarian and fallopian tubal cancer: FIGO stage I-IIIB
* Patients who undergoing surgery including pelvic and/or para-aortic lymph node dissection
* Patients with adequate bone marrow, renal and hepatic function:

WBC > 3,000 cells/mcl Platelets >100,000/mcl Creatinine <2.0 mg/dL Bilirubin <1.5 x normal and SGOT or SGPT <3 x normal

* American Society of Anesthesiology Physical Status 0-1
* Performance status of ECOG 0-2
* Patient must be suitable candidates for surgery
* Patients who have signed an approved Informed Consent

Exclusion Criteria:

* Patients with a history of pelvic or abdominal radiotherapy;
* Patients who are pregnant
* Patients with contraindications to surgery;
* Patients who are unfit for Surgery: serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator);
* Patient's compliance and geographic proximity that do not allow adequate follow-up.
* Patients who undergo only lymph node sampling

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Incidence of lymphocele an lymphatic ascites | within 1 year after surgery

SECONDARY OUTCOMES:
Time interval from surgery to removal of closed drain system | with 2 weeks after surgery
Postoperative drain amount | with 2 weeks after surgery
Postoperative hospital stay | within 2 weeks after surgery
Postoperative bleeding incidence | within 2 weeks after surgery
Postoperative complication incidence | within 1 month after surgery
Quality of life | within 1 year after surgery
2-year disease free survival and overall survival | 2 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Hyun Nam, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea